CLINICAL TRIAL: NCT00958750
Title: Investigator-initiated Single Blind, Two-armed, Randomized Phase 3 Clinical Trial to Compare Efficacy of 5% Minoxidil Topical Foam (5% Mtf) Once Daily Versus 2% Minoxidil Topical Solution (2% Mts) Twice Daily in Application on Females With Slightly to Moderate Androgenetic Alopecia Concerning Hair Volume
Brief Title: Efficacy and Safety Study to Compare Two Minoxidil Formulations on Women With Androgenetic Alopecia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Ulrike Blume-Peytavi, Clinical Research Center for Hair and Skin Science, Charité-Universitaetsmedizin Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRC-AGA01; EudraCT: 2008-001770-33
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2009-08

CONDITIONS: Androgenetic Alopecia; Female Pattern Hair Loss
Keywords: Androgenetic alopecia; female pattern hair loss
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5% MTF (Active Comparator): 5% minoxidil topical foam used once daily
  Interventions: Drug: minoxidil
- 2% MTS (Active Comparator): 2% minoxidil topical solution twice daily use
  Interventions: Drug: minoxidil

INTERVENTIONS:
Drug: minoxidil — the investigators compared two different formulations and concentrations of minoxidil in this study

SUMMARY:
The purpose of this study is to determine in women the risk/benefit profile and non-inferiority of a topical 5% Minoxidil foam formulation applied once daily for the treatment of androgenetic alopecia in comparison to 2% MTS used twice daily, using objective and subjective efficacy measures and safety assessments for a study period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 or older, in general good health
* Exhibits AGA based on a discernable decrease in hair density on the top of the scalp, relative to the sides and back of the scalp, with scalp hair density in involved area D3 to D6 on the Savin Density Scale (See Appendix 1)
* Hair density equal or less than 220 hairs /cm2 measured with TrichoScan
* Subjects who give their consent to the study after thoroughly clarification and who personally signed and dated the informed consent document indicating that the subject (or a legally acceptable representative), has been informed of all pertinent aspects of the trial
* Women of childbearing potential, who practice an effective method of contraception for at least five consecutive weeks prior to the study entry and during the study with one of the following methods:
* Double contraceptive method among hormonal contraception (e.g. contraceptive pill, intra uterine device, vaginal ring, injectable or implantable contraception), spermicide, condom and diaphragm. Oral/systemic contraception must have been the same during the past 6 months and will not be changed during the study
* Sexual abstinence
* Partner with a vasectomy (dated back more than 6 months) OR
* Women of non-childbearing potential, i. e. postmenopausal (absence of menstrual bleeding for 2 years), or had hysterectomy, bilateral tubal ligation or bilateral ovariectomy
* Women of childbearing potential must show a negative urine pregnancy test at Screening
* Willing to maintain the same hairstyle, hair length and hair color throughout the study
* Subjects who are willing and able to comply with scheduled visits, treatment plan, mini-tattoo, laboratory test and other trial procedures.

Exclusion Criteria:

* Known to be hypersensitive to Minoxidil, hair dye (P-Phenylendiamin), Tattoo ink, propylene glycol, fragrances, hair gel or any vehicle components.
* Current or 4 weeks dated back use of local treatment (drug or cosmetically) in the target region interfering with the study product or examination method (corticosteroids, Aminexil, Minoxidil, medical shampoos, topical estrogen, Ketoconazol)
* Current or 3 months dated back use of systemic treatment (drugs or dietary supplement) taken for more than 2 consecutive weeks interfering with the study product or examination method (beta blocker, Cimetidine, Diazoxid, Isotretinoin, corticosteroids, vitamin A intake above 10000 IU per day)
* Within past 6 month receiving of chemotherapy/cytotoxic agents as well as radiation and/or laser/surgical therapy of the scalp
* Current or prior enrollment in any other investigational medication (drug) study within the last 4 weeks
* Women with childbearing potential and insufficient contraception.
* Female who is pregnant, planning a pregnancy (during the course of the study) or nursing a child
* Presence of hair transplants, hair weaves or non-breathable wigs
* Any dermatological disorders of the scalp in the target region with the possibility of interfering with the study product or examination method, such as fungal or bacterial infections, seborrheic dermatitis, psoriasis, eczema, folliculitis, scars or scalp atrophy
* Active hair loss or history within the past 3 months including diffuse telogen effluvium, alopecia areata, scarring alopecia and androgen hair loss /hyper-androgenemia)
* Other severe, acute or chronic medical condition that may lead to hair loss or interfere with the interpretation of trial results
* Individuals who are institutionalized by court or regulatory order

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change of target area non-vellus hair count (TAHC) [n/cm²] after 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Assessing the investigational products safety by means of clinical examination (local intolerance, facial hypertrichosis, AE, SAE) and blood Minoxidil level (baseline + week 24) | 24 weeks
Change of cumulative hair width in non-vellus hair (TAHW) after 24 weeks | 24 weeks
Global expert panel rating of change in scalp coverage via assessment of global photographs | 24 weeks
Volunteer questionnaire rating for administration and contentment of the study product | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charité-Universitaetsmedizin; Clinical Research Center for Hair and Skin Science, Berlin, Germany